CLINICAL TRIAL: NCT02939599
Title: Long-term, Open Label, Multicenter, Extension Study to Evaluate the Safety and Tolerability of QCC374 in Patients With Pulmonary Arterial Hypertension (PAH)
Brief Title: Long-term Extension Study of the Safety and Pharmacokinetics of QCC374 in PAH Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated early for strategic reasons. Only Part I of the study was completed.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CQCC374X2201E1
Record Dates: First submitted 2016-10-12; First posted 2016-10-20 (Estimated); Results first posted 2020-02-28 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-02

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary hypertension (PH),; Increase blood pressure in the pulmonary artery; Increased blood pressure in the pulmonary vein; Increased blood pressure in the lung vasculature; Shortness of breath; Dizziness; Fainting; Leg swelling; Cough; Angina pector
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary; Dyspnea; Dizziness; Syncope; Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- QCC374 (Experimental): placebo patients from QCC374X2201 rolled into extension study will start at 0.03mg b.i.d. or 0.06mg b.i.d. and have the opportunity to up-titrate 0.12mg
  -active patients will continue at the dose they finished on the QCC374X2201 study
  Interventions: Drug: QCC374

INTERVENTIONS:
Drug: QCC374 — 0.015mg and 0.06mg

SUMMARY:
This is a long-term open-label safety extension to the Phase 2a study of inhaled QCC374 in adult patients with PAH. This study provides the patients who completed the QCC374X2201 study with the option to continue receiving QCC374. The study will monitor the long-term safety, tolerability and efficacy of QCC374 in patients with PAH.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.
* Subject was enrolled in the QCC374X2201 study and completed per protocol

Exclusion Criteria:

* Subjects who have started receiving prostacyclin (epoprostenol), prostacyclin analogs (i.e. trepostinil, iloprost, beraprost) or prostacyclin receptor agonists (i.e. selexipag) since the last study drug intake in the QCC374X2201 study.
* Females who are pregnant, or who plan to become pregnant during the study, or who are breastfeeding
* Any known factor or disease that may interfere with treatment compliance or study conduct (i.e. drug or alcohol dependence)
* Subjects who withdrew consent from the study QCC374X2201

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-11-06 (Actual); Study Completion 2018-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Novartis Investigative Site, Pittsburgh, Pennsylvania, United States
- Germany (2):
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Heidelberg
- Novartis Investigative Site, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=486

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Subjects randomized in the QCC374X2201 core study continued on QCC374 at their highest stable dose, in this extension study
- Arm 2: Subjects randomized to placebo in the QCC374X2201 core study completed a titration scheme similar to that of the active arm in QCC374X2201 core study protocol
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 3 | 2
Completed | 0 | 0
Not Completed | 3 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Study Terminated By Sponsor | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Subjects randomized in the QCC374X2201 core study continued on QCC374 at their highest stable dose, in this extension study 0.12mg
  -active patients will continue at the dose they finished on the QCC374X2201 study
- Arm2: Subjects randomized to placebo in the QCC374X2201 core study completed a titration scheme similar to that of the active arm in QCC374X2201 core study protocol
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm2 | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.3 (4.93) | 58.0 (9.90) | 47.4 (11.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Adverse Events (AEs), Serious Adverse Events (SAEs) in Patients With PAH Over a Two Year Period
Description: Patients with all (serious and non-serious) adverse events, serious adverse events and death were reported
Time Frame: Two years
Population: Safety set includes all participants who received at least one dose of study drug
Measure: Number; unit: Participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 3 | 2
Participants
  Participant with AE | 2 | 2
  Participants with serious AE | 1 | 0

2. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Cmax is the maximum (peak) observed plasma drug concentration after single dose administration. PK parameters were calculated from plasma concentration-time data using non-compartmental methods. Only descriptive analysis performed
Time Frame: 16 weeks
Population: Participants from the Pharmacokinetic (PK) analysis set, defined as all randomized participants who received at least one dose of study drug and one evaluable PK concentration measurement, with data available for analysis were considered
Measure: Median (Full Range); unit: pg/mL
Arm/Group | QCC374
Number analyzed (Participants) | 1
pg/mL
  QCC374: Day 1, Dose Level 0.03 mg | 82 [82 to 82]
  QCC374: Day 112, Dose Level 0.12 mg | 664 [664 to 664]

3. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax)
Description: Tmax is the time to reach maximum plasma concentration after single dose administration. PK parameters were calculated from plasma concentration-time data using non-compartmental methods. Only descriptive analysis performed.
Time Frame: 16 Weeks
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | QCC374
Number analyzed (Participants) | 1
hour
  QCC374: Day 1, Dose Level 0.03 mg | 0.250 [0.250 to 0.250]
  QCC374: Day 112, Dose Level 0.12 mg | 0.0330 [0.0330 to 0.0330]

4. Secondary Outcome: Area Under the Plasma Concentration-time Curve From 0 to the Last Measurable Concentration (AUClast)
Description: AUClast is the area under the plasma concentration-time curve from time zero to the last measurable concentration sampling time. PK parameters were calculated from plasma concentration-time data using non-compartmental methods. Only descriptive analysis performed.
Time Frame: 16 weeks
Population: as for outcome 2
Measure: Median (Full Range); unit: h*pg/mL
Arm/Group | QCC374
Number analyzed (Participants) | 1
h*pg/mL
  QCC374: Day 1, Dose Level 0.03 mg | 118 [118 to 118]
  QCC374: Day 112, Dose Level 0.12 mg | 526 [526 to 526]

5. Secondary Outcome: Area Under the Plasma Concentration Time Curve From 0 to the End of a Dosing Interval (AUCtau)
Description: AUCtau is the area under the plasma concentration-time curve from time zero to the end of the dosing interval. PK parameters were calculated from plasma concentration-time data using non-compartmental methods. Only descriptive analysis performed
Time Frame: 16 Weeks
Population: as for outcome 2
Measure: Median (Full Range); unit: h*pg/mL
Arm/Group | QCC374
Number analyzed (Participants) | 1
h*pg/mL
  QCC374: Day 1, Dose Level 0.03 mg | 134 [134 to 134]
  QCC374: Day 112, Dose Level 0.12 mg | 566 [566 to 566]

6. Secondary Outcome: Change From Baseline in Six Minute Walk Distance (6MWD)
Description: The Six Minute Walk Test measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is able to self-pace and rest as needed as they traverse back and forth along a marked walkway. Only descriptive analysis performed.
Time Frame: 16 weeks
Population: Participants from the Pharmacodynamic (PD) analysis set, defined as all randomized participants who received at least one dose of study drug and one evaluable PD assessment, with data available for analysis were considered.
Measure: Mean (Standard Deviation); unit: Meter
Arm/Group | QCC374
Number analyzed (Participants) | 3
Meter | 452 (104.65)

7. Secondary Outcome: Change in Tricuspid Annular Peak Systolic Velocity (TA S') at Week 16 (Day 112) Using Echocardiography
Description: Key Right Ventricular (RV) function endpoints such as Tricuspid Annular Peak Systolic Velocity (TA S') were assessed with echocardiography. Only descriptive analysis performed.
Time Frame: Two Years
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | QCC374
Number analyzed (Participants) | 1
cm/s | 10.90 (NA) — NA: Not estimable due to insufficient number of participants

8. Secondary Outcome: Change From Baseline in RV Tei Index at Week 16 (Day 112) Using Echocardiography
Description: Key Right Ventricular (RV) function endpoints such as Tei Index were assessed with echocardiography. The RV Tei index is using both systolic and diastolic time intervals to evaluate the overall global dysfunction of the right ventricle in PAH patients. A lower number in RV Tei Index indicates an improvement. Only descriptive analysis performed.
Time Frame: 16 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | QCC374
Number analyzed (Participants) | 1
Index | 0.84 (NA) — NA: Not estimable due to insufficient number of participants

9. Secondary Outcome: Change From Baseline in RV Fractional Area Change at Week 16 (Day 112) Using Echocardiography
Description: as for outcome 8
Time Frame: 16 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | QCC374
Number analyzed (Participants) | 1
Percentage change | 23.91 (NA) — NA: Not estimable due to insufficient number of participants

ADVERSE EVENTS:
Time Frame: through study completion an average of 4.5 months
Groups:
- QCC374 Arm 1: Subjects randomized in the QCC374X2201 core study continued on QCC374 at their highest stable dose, in this extension study 0.12mg -active patients will continue at the dose they finished on the QCC374X2201 study
- QCC374 Arm 2: Subjects randomized to placebo in the QCC374X2201 core study completed a titration scheme similar to that of the active arm in QCC374X2201 core study protocol
Arm/Group | QCC374 Arm 1 | QCC374 Arm 2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/2
Other Adverse Events (participants affected / at risk) | 1/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QCC374 Arm 1 (N=3) | QCC374 Arm 2 (N=2)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QCC374 Arm 1 (N=3) | QCC374 Arm 2 (N=2)
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2
Sunburn (Injury, poisoning and procedural complications) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 2
Headache (Nervous system disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/99/NCT02939599/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-04): https://cdn.clinicaltrials.gov/large-docs/99/NCT02939599/SAP_001.pdf